CLINICAL TRIAL: NCT03674450
Title: A Pilot Study at a Single Institution of Heart Rate Variability Biofeedback on Lung Cancer Patients Receiving Radiation Thearpy
Brief Title: Lung Heart Rate Variability
Acronym: HRV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study never enrolled any subjects. It was terminated due to staffing and technology changes.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 05518
Record Dates: First submitted 2018-09-10; First posted 2018-09-17 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental)
  Interventions: Behavioral: Heart Rate Variability Biofeedback Training

INTERVENTIONS:
Behavioral: Heart Rate Variability Biofeedback Training — The study will utilize the Physiolab GP8 heart rate variability and respiration system on a laptop computer used solely for the study with the proper security passwords to protect participant information. The equipment consists of two electrocardiogram sensors (one per wrist) attached by sports wrist bands, a respiration monitoring belt placed around the upper abdomen, two galvanic skin conductance sensors attached to the fingertips, and a thermistor sensor attached to one of the finger tips. Participants will perform a series of monitored breathing exercises.

SUMMARY:
The purpose of this study is to examine the effects of heart-rate variability biofeedback training on lung cancer patients receiving definitive radiation therapy. The target population consists of non-small cell lung cancer (NSCLC) patients receiving 6 weeks of radiation therapy. The study will utilize the Physiolab GP8 heart rate variability and respiration system to collect data as well as several survey instruments to analyze quality of life measures. The goal is to show the HRV training can improve certain QOL measures like anxiety and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be older than 18 years of age
* Both women and men of all ethnic background are eligible to participate in the study.
* Must be diagnosed with non-small cell lung cancer and receiving 6 weeks of radiation therapy.
* Must be available and willing to participate in 4, approximately 1 hour HRV biofeedback treatment sessions.
* Signed informed consent

Exclusion Criteria:

* Participant is younger than 18 or older than 70
* Diagnosed with early stage NSCLC
* Patients who are pregnant
* Patients with cardiac arrhythmias
* Patients with Pacemakers
* Patients taking beta-blockers
* Patients with any major mental illness, cognitive impairment
* Incapable of giving informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
EORTC QLQ-C30 Questionnaire | 2 years
  Questionnaire developed to assess the quality of life of cancer patients. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 2 years
  Measure the quality and patterns of sleep in adults. It differentiates from "poor" and "good" sleep quality by measuring seven areas. The order of the PSQI items has been modified from the original order in order to fit the first 9 items (which are the only items that contribute to the total score). Item 10 does not contribute to the PSQI score. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: William Levin, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ancoli-Israel S, Moore PJ, Jones V. The relationship between fatigue and sleep in cancer patients: a review. Eur J Cancer Care (Engl). 2001 Dec;10(4):245-55. doi: 10.1046/j.1365-2354.2001.00263.x. PMID 11806675
- [Background] Badger TA, Braden CJ, Mishel MH, Longman A. Depression burden, psychological adjustment, and quality of life in women with breast cancer: patterns over time. Res Nurs Health. 2004 Feb;27(1):19-28. doi: 10.1002/nur.20002. PMID 14745853
- [Background] Guo Y, Koshy S, Hui D, Palmer JL, Shin K, Bozkurt M, Yusuf SW. Prognostic Value of Heart Rate Variability in Patients With Cancer. J Clin Neurophysiol. 2015 Dec;32(6):516-20. doi: 10.1097/WNP.0000000000000210. PMID 26629761
- [Background] Hassett AL, Radvanski DC, Vaschillo EG, Vaschillo B, Sigal LH, Karavidas MK, Buyske S, Lehrer PM. A pilot study of the efficacy of heart rate variability (HRV) biofeedback in patients with fibromyalgia. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):1-10. doi: 10.1007/s10484-006-9028-0. Epub 2007 Jan 12. PMID 17219062
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Karavidas MK, Lehrer PM, Vaschillo E, Vaschillo B, Marin H, Buyske S, Malinovsky I, Radvanski D, Hassett A. Preliminary results of an open label study of heart rate variability biofeedback for the treatment of major depression. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):19-30. doi: 10.1007/s10484-006-9029-z. Epub 2007 Mar 1. PMID 17333315
- [Background] Liu L, Ancoli-Israel S. Sleep Disturbances in Cancer. Psychiatr Ann. 2008 Sep 1;38(9):627-634. doi: 10.3928/00485713-20080901-01. No abstract available. PMID 21243092
- [Background] Reiner R. Integrating a portable biofeedback device into clinical practice for patients with anxiety disorders: results of a pilot study. Appl Psychophysiol Biofeedback. 2008 Mar;33(1):55-61. doi: 10.1007/s10484-007-9046-6. Epub 2008 Feb 20. PMID 18286369